CLINICAL TRIAL: NCT06066515
Title: A Phase 3, Randomised, Double-blind, Parallel-group, 76-week, Efficacy and Safety Study of BI 456906 Administered Subcutaneously Compared With Placebo in Participants With Overweight or Obesity Without Type 2 Diabetes
Brief Title: A Study to Test Whether Survodutide (BI 456906) Helps People Living With Overweight or Obesity Who do Not Have Diabetes to Lose Weight
Acronym: SYNCHRONIZE™-1
Status: Active, not recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Boehringer Ingelheim (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 1404-0038; U1111-1288-9400 (Registry Identifier: WHO registry); 2022-502529-17-00 (Registry Identifier: CTIS)
Record Dates: First submitted 2023-09-27; First posted 2023-10-04 (Actual); Last update posted 2026-02-05 (Actual); Status verified 2026-02

CONDITIONS: Obesity
MeSH Terms: conditions — Obesity | interventions — BI 456906

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Survodutide 3.6 mg (Experimental)
  Interventions: Drug: survodutide
- Survodutide 6.0 mg (Experimental)
  Interventions: Drug: survodutide
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: survodutide — once weekly subcutaneous injection
  Other Names: BI 456906
  Arms: Survodutide 3.6 mg; Survodutide 6.0 mg
Drug: Placebo — once weekly subcutaneous injection
  Arms: Placebo

SUMMARY:
This study is open to adults who are at least 18 years old and have

* a body mass index (BMI) of 30 kg/m² or more, or
* a BMI of 27 kg/m² or more and at least one health problem related to their weight.

People with type 2 diabetes cannot take part in this study. Only people who have previously not managed to lose weight by changing their diet can participate.

The purpose of this study is to find out whether a medicine called survodutide (BI 456906) helps people living with overweight or obesity to lose weight. Participants are divided into 3 groups by chance, like drawing names from a hat. 2 groups get different doses of survodutide and 1 group gets placebo. Placebo looks like survodutide but does not contain any medicine. Every participant has a 2 in 3 chance of getting survodutide. Participants inject survodutide or placebo under their skin once a week for about one and a half years. In addition to the study medicine, all participants receive counselling to make changes to their diet and to exercise regularly.

Participants are in the study for about 1 year and 7 months. During this time, it is planned that participants visit the study site up to 14 times and receive 6 phone calls by the site staff.

The doctors check participants' health and take note of any unwanted effects. The participants' body weight is regularly measured. The results are compared between the groups to see whether the treatment works.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female, age ≥18 years at the time of signing informed consent, and at least the legal age of consent in countries where it is >18 years
2. Body mass index (BMI) ≥30 kg/m^2 at screening, OR BMI ≥27 kg/m^2 with the presence of at least one of the obesity-related complications (treated or untreated) e.g,:

   * Hypertension (defined as repeated, i.e. at least 3 measurements in resting condition, systolic blood pressure (SBP) values of ≥140 millimetre of mercury (mmHg) and/or diastolic blood pressure (DBP) values of ≥90 mmHg in the absence of anti-hypertensive treatment, or intake of at least 1 anti-hypertensive drug to maintain a normotensive blood pressure)
   * Dyslipidaemia (defined as at least 1 lipid-lowering treatment required to maintain normal blood lipid levels, or low-density lipoprotein (LDL) cholesterol ≥160 mg/dL (≥4.1 mmol/L), or triglycerides ≥150 mg/dL (≥1.7 mmol/L), or high-density lipoprotein (HDL) cholesterol <40 mg/dL (<1.0 mmol/L) for men or HDL cholesterol 50 mg/dL (<1.3 mmol/L) for women)
   * Obstructive sleep apnoea
   * Others.
3. History of at least one self-reported unsuccessful dietary effort to lose body weight.

Further inclusion criteria apply.

Exclusion Criteria:

1. Body weight change (self-reported) of >5% within 3 months before screening.
2. Treatment with any medication for the indication obesity within 3 months before screening.
3. Glycosylated haemoglobin A1c (HbA1c) ≥6.5% (≥48 mmol/mol) as measured by the central laboratory at screening.
4. History of type 1 diabetes mellitus (T1DM) or type 2 diabetes mellitus (T2DM) or treatment with glucose lowering agent started within 3 months before the screening up to and including the randomisation visit.
5. Heart failure (HF) with New York Heart Association (NYHA) functional class IV.
6. Known clinically significant gastric emptying abnormality (e.g. severe diabetic gastroparesis or gastric outlet obstruction).
7. History of either chronic or acute pancreatitis or elevation of serum lipase or serum pancreatic amylase >2x upper limit of normal (ULN) as measured by the central laboratory at screening.
8. Personal or family history of medullary thyroid carcinoma (MTC) or multiple endocrine neoplasia syndrome type 2 (MEN 2).

Further exclusion criteria apply.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 726 (Actual)
Dates: Start 2023-11-25 (Actual); Primary Completion 2025-10-28 (Actual); Study Completion 2026-02-13 (Estimated)

PRIMARY OUTCOMES:
Percentage change in body weight from baseline to Week 76 | Baseline and at Week 76
Achievement of body weight reduction ≥5% (yes/no) from baseline to Week 76 | Baseline and at Week 76

SECONDARY OUTCOMES:
Achievement of body weight reduction ≥10% (yes/no) from baseline to Week 76 | Baseline and at Week 76
Achievement of body weight reduction ≥15% (yes/no) from baseline to Week 76 | Baseline and at Week 76
Achievement of body weight reduction ≥20% (yes/no) from baseline to Week 76 | Baseline and at Week 76
Absolute change from baseline to Week 76 in body weight (kg) | Baseline and Week 76
Absolute change from baseline to Week 76 in waist circumference (cm) | Baseline and at Week 76
Absolute change from baseline to Week 76 in systolic blood pressure (SBP) (mmHg) | Baseline and at Week 76
Absolute change from baseline to Week 76 in "Capacity to Resist" domain score of the Eating Behaviour patient reported outcome (PRO) | Baseline and at Week 76
  "Capacity to Resist" domain score of the Eating Behaviour PRO is ranging between 0 and 24 and a higher score indicates a lower capacity to resist.
Absolute change from baseline to Week 76 in Eating Behaviour PRO total score | Baseline and at Week 76
  Eating Behaviour PRO total score is ranging between 0 and 48 and a higher score indicates a worse eating behaviour (greater desire to eat and/or lower capacity to resist).
Absolute change from baseline to Week 76 in body mass index (BMI) (kg/m2) | Baseline and at Week 76
Absolute change from baseline to Week 76 in diastolic blood pressure (DBP) (mmHg) | Baseline and at Week 76
Absolute change from baseline to Week 76 in glycosylated haemoglobin A1c (HbA1c) (%) | Baseline and at Week 76
Absolute change from baseline to Week 76 in HbA1c (mmol/mol) | Baseline and at Week 76
Absolute change from baseline to Week 76 in fasting plasma glucose (FPG) (mg/dL) | Baseline and at Week 76
Absolute change from baseline to Week 76 in fasting plasma insulin (FPI) (mIU/L) | Baseline and at Week 76
Absolute change from baseline to Week 76 in total cholesterol (mg/dL) | Baseline and at Week 76
Absolute change from baseline to Week 76 in high density lipoprotein (HDL) cholesterol (mg/dL) | Baseline and at Week 76
Absolute change from baseline to Week 76 in low density lipoprotein (LDL) cholesterol (mg/dL) | Baseline and at Week 76
Absolute change from baseline to Week 76 in very-low-density lipoprotein (VLDL) cholesterol (mg/dL) | Baseline and at Week 76
Absolute change from baseline to Week 76 in triglycerides (mg/dL) | Baseline and at Week 76
Absolute change from baseline to Week 76 in free fatty acids (mg/dL) | Baseline and at Week 76
Absolute change from baseline to Week 76 in alanine aminotransferase (ALT) (U/L) | Baseline and at Week 76
Absolute change from baseline to Week 76 in aspartate aminotransferase (AST) (U/L) | Baseline and at Week 76
Absolute change from baseline to Week 76 in total fat volume (L) | Baseline and at Week 76
Absolute change from baseline to Week 76 in lean body volume (L) | Baseline and at Week 76
Absolute change from baseline to Week 76 in visceral fat volume (L) | Baseline and at Week 76
Absolute change from baseline to Week 76 in subcutaneous fat volume (L) | Baseline and at Week 76.
Relative change from baseline to Week 76 in total fat volume (%) | Baseline and at Week 76
Relative change from baseline to Week 76 in lean body volume (%) | Baseline and at Week 76
Relative change from baseline to Week 76 in visceral fat volume (%) | Baseline and at Week 76
Relative change from baseline to Week 76 in subcutaneous fat volume (%) | Baseline and at Week 76.
Relative change from baseline to Week 76 in liver fat content (%) | Baseline and at Week 76

CONTACTS AND LOCATIONS:
Locations (118):
- United States (32):
  - EmVenio Research-Phoenix-69743, Phoenix, Arizona
  - Encompass Clinical Research, Spring Valley, Spring Valley, California
  - Diablo Clinical Research, Walnut Creek, California
  - Yale University School of Medicine, New Haven, Connecticut
  - Alliance for Multispecialty Research, LLC - Doral, Doral, Florida
  - University of Florida, Gainesville, Florida
  - East Coast Institute for Research, LLC - Jacksonville, Jacksonville, Florida
  - New Horizon Research Center-Miami-69732, Miami, Florida
  - West Orange Endocrinology, Ocoee, Florida
  - East-West Medical Research, Honolulu, Hawaii
  - Solaris Clinical Research, Meridian, Idaho
  - Evanston Premier Healthcare Research LLC, Skokie, Illinois
  - Velocity Clinical Research-Valparaiso-68883, Valparaiso, Indiana
  - Velocity Clinical Research-Sioux City-69728, Sioux City, Iowa
  - AMR Lexington, Lexington, Kentucky
  - L-MARC Research Center, Louisville, Kentucky
  - StudyMetrix Research, LLC, City of Saint Peters, Missouri
  - Premier Research, Inc., Trenton, New Jersey
  - Velocity Clinical Research - Binghamton, Binghamton, New York
  - Southgate Medical Group/ Southgate Medical Park, West Seneca, New York
  - Physicians East, PA, Greenville, North Carolina
  - Lucas Research, Inc., Morehead City, North Carolina
  - Accellacare-Wilmington-67123, Wilmington, North Carolina
  - Valley Weight Loss Clinic, Fargo, North Dakota
  - EmVenio Research-Oklahoma City-70053, Oklahoma City, Oklahoma
  - Trial Management Associates, Myrtle Beach, South Carolina
  - Texas Diabetes and Endocrinology, Austin, Texas
  - Juno Research, LLC, Houston, Texas
  - Diabetes & Glandular Disease Clinic, P.A., San Antonio, Texas
  - Consano Clinical Research, Shavano Park, Texas
  - Manassas Clinical Research Center, Manassas, Virginia
  - Rainier Clinical Research Center, Renton, Washington
- Australia (7):
  - Hunter Diabetes Centre, Merewether, New South Wales
  - CORE Research Group, Milton, Queensland
  - Griffith Health, Southport, Queensland
  - Monash University, Box Hill, Victoria
  - Austin Health, Heidelberg, Victoria
  - Baker Heart and Diabetes Institute, Melbourne, Victoria
  - Keogh Institute for Medical Research, Nedlands, Western Australia
- Belgium (4):
  - ASZ - Campus Aalst, Aalst
  - Edegem - UNIV UZ Antwerpen, Edegem
  - UZ Leuven, Leuven
  - Roeselare - HOSP AZ Delta, Roeselare
- Canada (10):
  - Dr. James Lai, Vancouver, British Columbia
  - Aggarwal and Associates Ltd., Brampton, Ontario
  - The Wharton Medical Clinic Clinical Trials Inc., Hamilton, Ontario
  - Milestone Research Inc., London, Ontario
  - James Cha, MD, Oshawa, Ontario
  - Stouffville Medical Research Institute Inc., Stouffville, Ontario
  - Albion Finch Medical Centre, Toronto, Ontario
  - Sameh Fikry Medicine Professional Corporation, Waterloo, Ontario
  - ViaCar Recherches Cliniques Inc. (Greenfield Park), Greenfield Park, Quebec
  - Power Clinical Research, Montreal, Quebec
- China (19):
  - Peking University People's Hospital, Beijing
  - Beijing Pinggu Hospital, Beijing
  - The First Hospital of Jilin University, Changchun
  - Changzhou Second People's Hospital, Changzhou
  - Guangdong Provincial People's Hospital, Guangzhou
  - Forth Clinical Hospital of Harbin Medical University, Harbin
  - Huzhou Central Hospital, Huzhou
  - Center Hospital of Jinan, Jinan
  - The First Affiliated Hospital of Henan University of Science and Technology, Luoyang
  - The Second Affiliated Hospital of Nanjing Medical University, Nanjing
  - Pingxiang People's Hospital, Pingxiang
  - Shanghai Municipal Hospital of Traditional Chinese Medicine, Shanghai
  - Shanghai Fifth People's Hospital affiliated to Fudan University, Shanghai
  - Siping Central People's Hospital, Siping
  - Suzhou Municipal Hospital, Suzhou
  - Tianjin Medical University General Hospital, Tianjin
  - The First Affiliated Hospital of Xi'an Medical University, Xi'an
  - The Second Affiliated Hospital of Zhengzhou University, Zhengzhou
  - Affiliated Hospital of Jiangsu University, Zhenjiang
- Finland (4):
  - HUS, Lihavuustutkimusyksikkö Biomedicum Helsinki, Helsinki
  - StudyCor Oy, Jyväskylä
  - Itä-Suomen yliopisto/Health Step Finland Oy, Kuopio
  - CRST - Clinical Research Services Turku, Turku
- Germany (4):
  - InnoDiab Forschung GmbH, Essen
  - MVZ im Altstadt-Caree Fulda GmbH, Fulda
  - Diabetes Zentrum Hamburg West, Hamburg
  - Institut für Diabetesforschung Münster GmbH, Münster
- Japan (5):
  - Fukuhama Chuo Clinic, Fukuoka, Fukuoka
  - Kobe University Hospital, Hyogo, Kobe
  - Noritake Clinic, Ibaraki, Ushiku
  - Soka Sugiura Naika Clinic, Saitama, Soka
  - Hachioji Diabetes Clinic, Tokyo, Hachioji
- Netherlands (3):
  - PT & R, Born
  - Universitair Medisch Centrum Groningen, Groningen
  - Franciscus Gasthuis, Rotterdam
- New Zealand (5):
  - P3 Research Dunedin, Dunedin
  - Southern Clinical Trials Tasman, Nelson
  - P3 Research-Newtown Wellington NZ-33770, Newtown Wellington NZ
  - Optimal Clinical Trials North, Rosedale, Auckland
  - P3 Research-Tauranga-34833, Tauranga
- Poland (5):
  - PI HOUSE Sp. z o.o., Gdansk, Gdansk
  - ETG Lublin, Lublin
  - Velocity Nova Sp z o.o., Puławy
  - ETG Siedlce, Siedlce
  - Clinical Research Center METABOLICA lek. Robert Witek, Tarnów
- South Korea (10):
  - The Catholic University of Korea, Bucheon St.Mary's Hospital, Bucheon-si
  - Kyungpook National University Hospital, Daegu
  - Dongguk University Ilsan Hospital, Goyang
  - Gachon University Gil Medical Center, Incheon
  - Seoul National University Bundang Hospital, Seongnam
  - Seoul National University Hospital, Seoul
  - Severance Hospital, Seoul
  - The Catholic University of Korea, Yeouido St.Mary's Hospital, Seoul
  - Kangbuk Samsung Hospital, Seoul
  - Ajou University Hospital, Suwon
- Sweden (4):
  - Ladulaas Kliniska Studier, Borås
  - Forskningsenheten Carlanderska, Gothenburg
  - Medicinmottagning 5/Överviktsenheten, Örebro
  - Sabbatsbergs sjukhus, Stockholm
- United Kingdom (6):
  - Waterloo Medical Centre, Blackpool
  - Bradford on Avon Health Centre, Bradford-on-Avon
  - Burbage Surgery, Burbage, Hinkley
  - Kiltearn Medical Centre, Nantwich
  - Clifton Medical Centre, Rotherham, Rotherham
  - Trowbridge Health Centre, Trowbridge

IPD SHARING:
Plan to Share IPD: Yes
Once the criteria in section 'time frame' are fulfilled, researchers can use the following link https:// www.mystudywindow.com/msw/datasharing to request access to the clinical study documents regarding this study, and upon a signed "Document Sharing Agreement". Furthermore, researchers can request access to the clinical study data, for this and other listed studies, after the submission of a research proposal and according to the terms outlined in the website.
Supporting Information: Study Protocol, SAP, CSR
Time Frame: After structured results have been posted, all regulatory activities are completed in the US and EU for the product and indication, and after the primary manuscript has been accepted for publication.
Access Criteria: For study documents - upon signing of a 'Document Sharing Agreement'.For study data -1. after the submission and approval of the research proposal (checks will be performed by the sponsor and/or the independent review panel, including checking that the planned analysis does not compete with sponsor's publication plan); 2. and upon signing of a legal agreement.
URL: https://www.mystudywindow.com/msw/datasharing

REFERENCES:
- [Derived] le Roux CW, Wharton S, Bozkurt B, Platz E, Bleckert G, Ajaz Hussain S, Brueckmann M, Startseva E, Kloer IM, Kaplan LM. Survodutide for treatment of obesity: Baseline characteristics of participants in a randomized, double-blind, placebo-controlled, phase 3 trial (SYNCHRONIZE-1). Diabetes Obes Metab. 2026 Jan;28(1):337-346. doi: 10.1111/dom.70196. Epub 2025 Nov 4. PMID 41187967
- See also: Related Info — http://www.mystudywindow.com